CLINICAL TRIAL: NCT01456000
Title: Pivotal Clinical Study of the CardioFocus Endoscopic Ablation System - Adaptive Contact (EAS-AC) or HEARTLIGHT for the Treatment of Symptomatic Atrial Fibrillation
Brief Title: HeartLight Ablation in Patients With Paroxysmal Atrial Fibrillation (PAF)
Acronym: HeartLight
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CardioFocus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-3002
Record Dates: First submitted 2011-10-17; First posted 2011-10-20 (Estimated); Results first posted 2016-09-08 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-07

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: atrial fibrillation; AF; PAF; PVI; ablation; paroxysmal atrial fibrillation; pulmonary vein isolation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EAS-AC (HeartLight) (Experimental): Treatment with the EAS-AC.
  Interventions: Device: EAS-AC (HeartLight)
- Control Arm Ablation (Active Comparator): Treatment with standard ablation.
  Interventions: Procedure: Control Arm Ablation

INTERVENTIONS:
Device: EAS-AC (HeartLight) — Pulmonary vien isolation
  Arms: EAS-AC (HeartLight)
Procedure: Control Arm Ablation — Treatment with standard ablation.
  Arms: Control Arm Ablation

SUMMARY:
The purpose of this study is to demonstrate the safety and effectiveness of the CardioFocus Endoscopic Ablation System with Adaptive Contact (HeartLight) in the treatment of atrial fibrillation by creating electrical isolation of the pulmonary veins.

DETAILED DESCRIPTION:
A randomized, controlled trial designed to demonstrate the safety and effectiveness of the experimental device to deliver pulmonary vein isolation as a treatment for symptomatic atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years.
* paroxysmal atrial fibrillation
* failure of at least one AAD
* others

Exclusion Criteria:

* overall good health as established by multiple criteria

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2012-01; Primary Completion 2014-12 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Burke Barrett, Study Director — CardioFocus, Inc. (sponsor); Vivek Reddy, MD, Principal Investigator — Mt. Sinai Hospital, NYC; Andrea Natale, MD, Principal Investigator — Texas Cardiac Arrhythmia Research Foundation
Locations (21):
- United States (21):
  - University of Alabama, Birmingham, Birminham, Alabama
  - Stanford Hospital, Palo Alto, California
  - Regional Cardiology Associates, Mercy General Hospital, Sacramento, California
  - UCSF, San Francisco, California
  - Pacific Heart Institute, Santa Monica, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Prairie Heart Institute, Springfield, Illinois
  - The University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beaumont Hospital, Royal Oak, Michigan
  - Mayo Clinic Rochester/St. Mary's Hospital, Rochester, Minnesota
  - Mt. Sinai Hospital, New York, New York
  - Duke University, Durham, North Carolina
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University South Carolina, Charleston, South Carolina
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - Methodist Hospital, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - Sentara Cardiovascular Research Institute, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dukkipati SR, Cuoco F, Kutinsky I, Aryana A, Bahnson TD, Lakkireddy D, Woollett I, Issa ZF, Natale A, Reddy VY; HeartLight Study Investigators. Pulmonary Vein Isolation Using the Visually Guided Laser Balloon: A Prospective, Multicenter, and Randomized Comparison to Standard Radiofrequency Ablation. J Am Coll Cardiol. 2015 Sep 22;66(12):1350-60. doi: 10.1016/j.jacc.2015.07.036. PMID 26383722

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 405 participants enrolled in the study. Thirty nine of these participants were enrolled in the run-in phase and are not reported in the pivotal data. Of the remaining 366 enrolled participants, 13 were excluded from the study prior to randomization, resulting in a total of 353 randomized participants.
Groups:
- EAS-AC (HeartLight): Treatment with the EAS-AC.
  EAS-AC (HeartLight): Pulmonary vien isolation
  ITT Population 178 participants
- Control Arm Ablation: Treatment with standard ablation.
  Control Arm Ablation: Treatment with standard ablation.
  ITT Population 175 Participants
Period: Overall Study
Arm/Group | EAS-AC (HeartLight) | Control Arm Ablation
Started | 178 | 175
Completed | 170 | 172
Not Completed | 8 | 3

BASELINE CHARACTERISTICS:
Population: Average Age
Groups:
- EAS-AC (HeartLight): Treatment with the EAS-AC. Randomized and treated cohort.
  EAS-AC (HeartLight): Pulmonary vien isolation
- Control Arm Ablation: Treatment with standard ablation. Randomized and treated cohort.
  Control Arm Ablation: Treatment with standard radiofrequency (RF) ablation.
- Total: Total of all reporting groups
Arm/Group | EAS-AC (HeartLight) | Control Arm Ablation | Total
Number analyzed (Participants) | 170 | 172 | 342
Age, Customized [Mean (Standard Deviation); unit: Years]
  Age | 59.7 (10.4) | 60.1 (8.9) | 59.9 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 63 | 115
  Male | 118 | 109 | 227
Region of Enrollment [Number; unit: participants]
  United States | 170 | 172 | 342

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Meeting the Efficacy Success Criteria as Described in the Outcome Measure Description
Description: Episodes of AF were monitored during the follow-up period and the rate of participants with no documented, symptomatic episodes of AF in follow-up were be compared. Other efficacy success/failure criteria included acute isolation of all clinically relevant pulmonary veins, lack of ablation-induced left atrial flutter, use of AADs during a follow-up period and left heart ablation or implant for AF in follow-up. Randomized and treated participants that were evaluable for efficacy are reported on for the Outcome Measure.
Time Frame: 1 year
Measure: Number; unit: Successful Participants
Groups:
- EAS-AC (HeartLight): Treatment with the EAS-AC and evaluable for efficacy.
  EAS-AC (HeartLight): Pulmonary vien isolation
- Control Arm Ablation: Treatment with standard ablation and evaluable for efficacy.
  Control Arm Ablation: Treatment with standard ablation.
Arm/Group | EAS-AC (HeartLight) | Control Arm Ablation
Number analyzed (Participants) | 167 | 167
Successful Participants | 102 | 103

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse event data were collected from the time of ablation (day 0) through 1 year of follow-up
Arm/Group | EAS-AC (HeartLight) | Control Arm Ablation
Serious Adverse Events (participants affected / at risk) | 16/170 | 10/172
Other Adverse Events (participants affected / at risk) | 92/170 | 105/172
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EAS-AC (HeartLight) (N=170) | Control Arm Ablation (N=172)
Cardiac perforation, pericardial effusion or tamponade (Cardiac disorders) | 3 (3) | 4 (4)
CVA or stroke (Nervous system disorders) | 1 (1) | 1 (1) — cerebrovascular event or stroke
Chest pain or pericarditis (Cardiac disorders) | 2 (2) | 4 (4)
Diaphragmatic paralysis or phrenic nerve injury (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0)
Hemorrhage or pseudoaneurysm (Vascular disorders) | 2 (2) | 0 (0)
Other (Cardiac disorders) | 3 (3) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EAS-AC (HeartLight) (N=170) | Control Arm Ablation (N=172)
Cardioversion (Cardiac disorders) | 14 (14) | 16 (16)
Chest pain/discomfort (Cardiac disorders) | 5 (5) | 11 (11)
Pericardial effusion (Cardiac disorders) | 8 (8) | 14 (14)
Other (Cardiac disorders) | 65 (65) | 64 (64) — All other events reported below the 5% reporting threshold.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No